CLINICAL TRIAL: NCT07200102
Title: Selinexor Maintenance Post CAR-T Cell Therapy for Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202511028
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Cilta-cel; Selinexor; Multiple Myeloma; Maintenance
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selinexor (Experimental): Patients with high risk of relapse will receive selinexor starting between Day 30 - Day 58 after cilta-cel infusion for up to 12 cycles (initiation of treatment may be delayed from day 30 for up to 28 days to allow for MRD testing to results or for a patient experiencing ongoing cytopenias). Selinexor will be given weekly on Days 1, 8, 15, and 22 of each 28-day cycle. The first 3 to 6 patients enrolled will be part of the safety run-in cohort; these patients will be monitored for dose-limiting toxicities during Cycle 1. Provided the safety run-in shows that selinexor is safe and tolerable at this dose, an additional 14 to 17 patients (for a total of 20) will be enrolled.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Selinexor will be provided by Karyopharm Therapeutics, Inc.
  Other Names: KPT-330; Xpovio

SUMMARY:
The outcomes in patients with relapsed multiple myeloma refractory to triple-therapy (anti-CD38, immunomodulatory drugs (IMiD) and proteasome inhibitors (PI)) remain poor. These patients are eligible for chimeric antigen receptor T-cells (CAR-T), which rely on redirecting autologous T-cells to clear myeloma cells by targeting B-cell maturation antigen (BCMA). BCMA CAR-T therapy is not curative, and unlike autologous stem cell transplant, there is currently no standard for maintenance therapy post CAR-T which could potentially increase MRD rates and extend progression-free survival.

Selinexor is an exportin (XPO1) inhibitor with direct anti-tumor effect used often as an adjunct with other agents as bridging therapy prior to CAR-T. As selinexor does not affect T-cell yields or fitness, T-cell collection on selinexor for CAR-T manufacturing is safe.

The aim of this study is to evaluate the safety and toxicity of selinexor in triple-exposed or refractory multiple myeloma patients with high-risk features (adverse risk cytogenetics, less than complete response (CR) post CAR-T, or extramedullary disease) following BCMA CAR-T therapy. The investigators hypothesize that selinexor as maintenance therapy following CAR-T has the potential to act synergistically with CAR-T cells leading to more durable responses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of triple-class exposed or refractory multiple myeloma. Diagnosis must be histologically confirmed. Patients with multiple myeloma with local amyloid deposition in the bone marrow are eligible.
* Received standard of care ciltacabtagene autoleucel (cilta-cel; Carvykti).
* High risk cytogenetics as defined by IMWG OR Presence of extramedullary disease documented prior to receiving CAR-T OR Patients with less than CR at Day 30 post CAR-T OR Patients with MRD-positive disease at Day 30 post CAR-T
* Able to monitor disease response by ClonoSEQ MRD testing.
* At least 18 years of age.
* ECOG performance status ≤ 2.
* Adequate bone marrow and organ function at Day 30 post CAR-T (+28 /-14 days) as defined below:

  * Absolute neutrophil count ≥ 1.0 K/cumm
  * Platelets ≥ 50 K/cumm
  * Hemoglobin ≥ 8.5 g/dL without blood transfusion within 7 days before C1D1.
  * Total bilirubin ≤ 1.5 x IULN; patients with Gilbert's syndrome must have a total bilirubin < 3 x IULN.
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Calculated creatinine clearance ≥ 15 mL/min by Cockcroft-Gault
* The effects of selinexor on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days after completion of selinexor. Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* MM with active CNS involvement.
* Confirmed progressive disease by IMWG after CAR-T administration.
* Unresolved cytokine release syndrome (CRS) or CAR-T neurologic toxicity.
* Any unresolved non-hematologic grade ≥ 3 treatment-related toxicity from CAR-T.
* Administration or planned administration of any other concomitant chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy which would be considered a treatment of multiple myeloma from Day 28 post-CAR-T cell therapy through discontinuation from study treatment. Note: patients may be on corticosteroids if they are being given for disorders other than multiple myeloma (e.g., adrenal insufficiency, rheumatoid arthritis)
* Has received selinexor or another XPO1 inhibitor post-CART.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Prior organ transplant requiring immunosuppressive therapy.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to selinexor or other agents used in the study.
* Active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to CAR-T (patients on prophylactic antibiotics or with a controlled infection within 1 week prior to CAR-T may enroll); active, unstable cardiovascular function, as indicated by the presence of symptomatic ischemia, uncontrolled clinically significant conduction abnormalities (e.g. patients with ventricular or atrial tachycardia on anti-arrhythmics are excluded; patients with first degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), congestive heart failure of NYHA class ≥ 3 or known left ventricular ejection fraction of < 40%, or myocardial infraction within 3 months prior to CAR-T therapy.
* Major surgery within 28 days prior to CAR-T cell therapy.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of study entry.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible. HIV testing not required in the absence of known history of infection.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible. HBV testing not required in the absence of known history of infection.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible. HCV testing not required in the absence of known history of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of non-hematologic grade ≥ 3 treatment-related adverse events (excluding conditioning and CAR-T related adverse events) according to CTCAE v 5.0 | From start of selinexor through 30 days after the last dose of selinexor (estimated to be 13 months)
Tolerability as measured by rate of patients who received > 80% of cumulative selinexor dose during the study period | Through completion of selinexor treatment (estimated to be 12 months)

SECONDARY OUTCOMES:
Rate of MRD negativity by clonoSEQ sensitive to 10-5 | At 6 months after CAR-T infusion
Rate of MRD negativity by clonoSEQ sensitive to 10-5 | At 12 months after CAR-T infusion
Rate of complete response (CR) and stringent CR (sCR) by IMWG response criteria | At 6 months after CAR-T infusion
  * sCR: Stringent complete response requires all of the following:
    * CR as defined below
    * Normal free light chain ratio (0.26-1.65)
    * Absence of clonal cells in the bone marrow by immunohistochemistry or immunofluorescence
  * CR: Complete response requires all of the following:
    * Negative immunofixation on the serum and urine
    * <5% plasma cells in the bone marrow aspirate
    * Disappearance of any soft tissue plasmacytomas
Rate of complete response (CR) and stringent CR (sCR) by IMWG response criteria | At 12 months after CAR-T infusion
  * sCR: Stringent complete response requires all of the following:
    * CR as defined below
    * Normal free light chain ratio (0.26-1.65)
    * Absence of clonal cells in the bone marrow by immunohistochemistry or immunofluorescence
  * CR: Complete response requires all of the following:
    * Negative immunofixation on the serum and urine
    * <5% plasma cells in the bone marrow aspirate
    * Disappearance of any soft tissue plasmacytomas
Progression-free survival (PFS) | At 6 months after CAR-T infusion
  PFS is defined as: The time from initiation of treatment to the occurrence of either objective disease progression (by IMWG criteria) or death from any cause, whichever comes first.
Progression-free survival (PFS) | At 12 months after CAR-T infusion
  PFS is defined as: The time from initiation of treatment to the occurrence of either objective disease progression (by IMWG criteria) or death from any cause, whichever comes first.
Time to progression (TTP) | Through completion of follow-up (estimated to be 24 months)
  TTP is defined as: The interval from initiation of therapy to the first documentation of disease progression, as determined by IMWG criteria.
Duration of response (DOR) | Through completion of follow-up (estimated to be 24 months)
  DOR is defined as: The time interval from the first documented evidence of a partial response or better after starting treatment by IMWG criteria to the occurrence of disease progression (by IMWG criteria) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Analysis will be performed to achieve the aims of the approved proposal.
  Contact the PI regarding proposal submission and accessing data.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu